CLINICAL TRIAL: NCT02659605
Title: Cord Clamping Level Above or Below Mother's Perineum
Acronym: CLAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Pamela Berens, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-11-0633
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Pre-term Birth; Delayed Cord Clamping
Keywords: pre-term birth; delayed cord clamping; skin to skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed cord clamping above the perineum (Experimental)
  Interventions: Procedure: Delayed cord clamping above the perineum
- Delayed cord clamping below the perineum (Active Comparator)
  Interventions: Procedure: Delayed cord clamping below the perineum

INTERVENTIONS:
Procedure: Delayed cord clamping above the perineum — After delivery, the infant will be placed on the mother's abdomen and the cord will be clamped 30-45 seconds after delivery of the infant.
  Arms: Delayed cord clamping above the perineum
Procedure: Delayed cord clamping below the perineum — The infant will be held below the perineum, and the cord clamped and cut 60-75 seconds after delivery of the infant.
  Arms: Delayed cord clamping below the perineum

SUMMARY:
The purpose of this study is to determine if delayed cord clamping above the perineum has an effect on neonatal hematocrit when compared to delayed cord clamping below the perineum in pre-term spontaneous vaginal deliveries.

DETAILED DESCRIPTION:
This study will compare the difference in neonatal hematocrit with delayed cord clamping above vs. below the perineum, in infants who are born via pre-term spontaneous vaginal deliveries that are vigorous at delivery. Delayed cord clamping below the perineum is an accepted clinical practice in obstetrics and gynecology; however, delayed cord clamping above the perineum has not yet been studied in preterm infants. Delayed cord clamping above the perineum will provide the benefit of immediate skin-to-skin contact between the mother and her newborn.

Patients will have delayed cord clamping performed for 60-75 seconds either below the maternal perineum or while the infant is placed on the mother's abdomen. At approximately 24 hours after delivery (at the time of infant heel stick for routine, state-mandated screening tests), a small additional amount of blood will be collected to evaluate newborn hematocrit.

ELIGIBILITY:
Inclusion Criteria:

* Singleton intrauterine pregnancies at least 30 weeks gestation but less than 37 weeks gestation

Exclusion Criteria:

* Acute febrile illnesses or chronic medical problems such as hypertension, diabetes mellitus, renal disease, medically-managed seizure disorders
* Pregnancy-related complications such as pre-eclampsia, intrauterine growth restriction, chromosomal/anatomical abnormalities, and placental abruption
* Infants who are not anticipated to undergo spontaneous vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Berens, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansaray A, Yetman R, Berens P. Effect of Delayed Cord Clamping Above Versus Below the Perineum on Neonatal Hematocrit: A Randomized Controlled Trial. Breastfeed Med. 2015 Dec;10(10):464-7. doi: 10.1089/bfm.2015.0109. PMID 26651542

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 subjects were consented, but 29 were determined to be ineligible prior to randomization (that is, 29 did not start the study).
Period: Overall Study
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
Started | 40 | 34
Completed | 31 | 30
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (6.0) | 26.8 (5.2) | 27.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 21 | 17 | 38
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 13 | 30
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 13 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 30 | 61
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  less than 25 kg/m^2 | 4 | 8 | 12
  greater than or equal to 25 kg/m^2 and below 30 kg | 9 | 7 | 16
  greater than or equal to 30 kg/m^2 | 18 | 15 | 33
Parity [Mean (Standard Deviation); unit: # previous pregnancies carried to term] | 1.7 (1.5) | 1.2 (1.2) | 1.4 (1.4)
Insurance [Count of Participants; unit: Participants]
  none/self-pay | 1 | 1 | 2
  Medicaid | 26 | 20 | 46
  private | 4 | 9 | 13
Prenatal care [Count of Participants; unit: Participants]
  prenatal care | 30 | 28 | 58
  no prenatal care | 1 | 2 | 3
Induced [Count of Participants; unit: Participants] | 20 | 19 | 39
Gestational age in weeks [Mean (Standard Deviation); unit: weeks] | 35.3 (1.2) | 34.6 (1.7) | 34.9 (1.7)
Gestational age greater than or equal to 32 weeks [Count of Participants; unit: Participants] | 31 | 26 | 57

OUTCOME MEASURES:

1. Primary Outcome: Hematocrit Level
Time Frame: 24 hours after delivery
Measure: Mean (Standard Deviation); unit: % of blood composed of red blood cells
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
Number analyzed (Participants) | 31 | 30
% of blood composed of red blood cells | 51.5 (8.4) | 52.6 (7.3)
Statistical Analysis 1: Comparison: Delayed Cord Clamping Above the Perineum vs Delayed Cord Clamping Below the Perineum; Test type: Equivalence — The sample size was based on a previous study by Rabe et al. (Obstet Gynecol. 2011;117(2 Pt 1):205-11), who were also evaluating neonatal hematocrit after delayed cord clamping with the intention of detecting a 10% difference with a p-value of 0.05 and a power of 80% for a two-sided t-test. That study determined that 26 patients in each group were needed for a total of 52 subjects; p = 0.572, Student's t-test

2. Secondary Outcome: Number of Participants With Infants Who Were Admitted to the Neonatal Intensive Care Unit (NICU)
Time Frame: during the initial hospital stay (1-2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
Number analyzed (Participants) | 31 | 30
Participants | 21 | 21
Statistical Analysis 1: Comparison: Delayed Cord Clamping Above the Perineum vs Delayed Cord Clamping Below the Perineum; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.849, Student's t-test

3. Secondary Outcome: Number of Participants With Infants Who Received Phototherapy
Time Frame: during the initial hospital stay (1-2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
Number analyzed (Participants) | 31 | 30
Participants | 14 | 13
Statistical Analysis 1: Comparison: Delayed Cord Clamping Above the Perineum vs Delayed Cord Clamping Below the Perineum; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.886, Student's t-test

4. Secondary Outcome: Number of Participants With Infants Who Received Blood Transfusion
Time Frame: during the initial hospital stay (1-2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
Number analyzed (Participants) | 31 | 30
Participants | 1 | 2
Statistical Analysis 1: Comparison: Delayed Cord Clamping Above the Perineum vs Delayed Cord Clamping Below the Perineum; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.612, Student's t-test

5. Secondary Outcome: Apgar Score at 1 Minute
Description: The Apgar score is a method to quickly summarize the health of newborn children. The Apgar score is determined by evaluating the newborn baby on five simple criteria (Appearance, Pulse, Grimace, Activity, Respiration) on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10, which zero associated with worse outcomes.
Time Frame: 1 minute after birth
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
Number analyzed (Participants) | 31 | 30
score | 7.8 (1.3) | 7.9 (1.5)
Statistical Analysis 1: Comparison: Delayed Cord Clamping Above the Perineum vs Delayed Cord Clamping Below the Perineum; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.728, Student's t-test

6. Secondary Outcome: Apgar Score at 5 Minutes
Description: as for outcome 5
Time Frame: 5 minutes after birth
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
Number analyzed (Participants) | 31 | 30
score | 8.7 (0.6) | 8.6 (0.9)
Statistical Analysis 1: Comparison: Delayed Cord Clamping Above the Perineum vs Delayed Cord Clamping Below the Perineum; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.584, Student's t-test

ADVERSE EVENTS:
Time Frame: during the initial hospital stay (1-2 days)
Arm/Group | Delayed Cord Clamping Above the Perineum | Delayed Cord Clamping Below the Perineum
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

LIMITATIONS AND CAVEATS:
Inability to blind participants and medical staff involved in the delivery. Data for some subjects was not obtained due to systems errors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02659605/Prot_000.pdf